CLINICAL TRIAL: NCT02160158
Title: Open-label, Single-dose, Randomized, Crossover Study To Estimate The Relative Bioavailability Compared To Commercial Extended-release Tablet Formulation And The Effects Of Food Or Sprinkling On Applesauce For Fesoterodine Sustained-release Beads-in-capsule Formulations In Healthy Adult Volunteers
Brief Title: Study to Estimate the Relative Bioavailability Compared to Commercial Extended-release Tablet Formulation and the Effects of Food Or Sprinkling on Applesauce for Fesoterodine Sustained-release Beads-in-capsule Formulations in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A0221099; 2014-001248-39 (EudraCT Number)
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Fesoterodine; SR3; SR4; bioavailability; pharmacokinetics; sprinkle; applesauce
MeSH Terms: interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: Fesoterodine ER (fasted); Drug: Fesoterodine SR3 (fasted); Drug: Fesoterodine SR3 (fed); Drug: Fesoterodine ER (fed); Drug: Fesoterodine SR3 (sprinkle)
- Cohort 2 (Experimental)
  Interventions: Drug: Fesoterodine ER (fasted); Drug: Fesoterodine SR4 (fasted); Drug: Fesoterodine SR4 (fed); Drug: Fesoterodine ER (fed); Drug: Fesoterodine SR4 (sprinkle)

INTERVENTIONS:
Drug: Fesoterodine ER (fasted) — Commercial Fesoterodine ER 4 mg (single dose)
  Arms: Cohort 1
Drug: Fesoterodine SR3 (fasted) — Fesoterodine SR3 4 mg (single dose)
  Arms: Cohort 1
Drug: Fesoterodine SR3 (fed) — Fesoterodine SR3 4 mg (single dose) with high-fat meal
  Arms: Cohort 1
Drug: Fesoterodine ER (fed) — Commercial Fesoterodine ER 4 mg (single dose) with high-fat meal
  Arms: Cohort 1
Drug: Fesoterodine SR3 (sprinkle) — Fesoterodine SR3 4 mg (single dose) beads sprinkled on applesauce
  Arms: Cohort 1
Drug: Fesoterodine ER (fasted) — Commercial Fesoterodine ER 4 mg (single dose)
  Arms: Cohort 2
Drug: Fesoterodine SR4 (fasted) — Fesoterodine SR4 4 mg (single dose)
  Arms: Cohort 2
Drug: Fesoterodine SR4 (fed) — Fesoterodine SR4 4 mg (single dose) with high-fat/high calorie meal
  Arms: Cohort 2
Drug: Fesoterodine ER (fed) — Commercial Fesoterodine ER 4 mg (single dose) with high-fat meal
  Arms: Cohort 2
Drug: Fesoterodine SR4 (sprinkle) — Fesoterodine SR4 4 mg (single dose) beads sprinkled on applesauce
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability of 2 new bead-in-capsule formulations compared to the commercial extended-release formulation (both fed and fasted) and to assess the effect of sprinkling the capsule contents on applesauce on the pharmacokinetics of 5 hydroxymethyl tolterodine (5-HMT).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years; Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication
* History of uncontrolled narrow angle glaucoma, myasthenia gravis, gastric retention, severe ulcerative colitis and toxic megacolon
* Evidence or history of clinically significant urologic disease [urinary retention, obstructive disturbance of bladder emptying, micturition disturbance, nocturia or pollacisuria (eg, benign prostate hyperplasia, urethral stricture, recurrent urinary tract infections); Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes/day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 48 hours
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Maximum Observed Plasma Concentration (Cmax) | 48 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 48 hours
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 48 hours
Plasma Decay Half-Life (t1/2) | 48 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221099&StudyName=Study%20to%20Estimate%20the%20Relative%20Bioavailability%20Compared%20to%20Commercial%20Extended-release%20Tablet%20Formulation%20and%20the%20Effects%20of%20Food%20Or%20Sprin